CLINICAL TRIAL: NCT07020273
Title: Cancer Prevention by Reducing Tobacco With Informatics and Chronic Care Approaches Trial (CONNECT)
Brief Title: CONNECT Cancer Survivors With Tobacco Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202503025
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use; Tobacco Use Cessation; Smoking Cessation; Nicotine Addiction; Tobacco Smoking
Keywords: Patient Reported Outcomes; Tobacco Treatment
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation; Smoking Cessation; Tobacco Use Disorder; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Randomization occurs at the clinic level. For pragmatic concerns, the investigators expect to recruit from multiple clinics and randomization will be stratified by department to minimize the clinic effect. Clinics will be randomized on a 1:1 basis to ELEVATE-S or ELEVATE. Patients within a clinic will be assigned to the same arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic health record-enabled evidence-based tobacco treatment (ELEVATE) (Active Comparator)
  Interventions: Behavioral: ELEVATE
- Electronic health record-enabled evidence-based tobacco treatment-Support (ELEVATE-S) (Experimental)
  Interventions: Behavioral: ELEVATE-S

INTERVENTIONS:
Behavioral: ELEVATE — ELEVATE uses implementation strategies to support clinicians (support clinicians by revising professional roles to enable point of care tobacco treatment with a team are approach and support clinicians by providing clinical decision support tools).
  Arms: Electronic health record-enabled evidence-based tobacco treatment (ELEVATE)
Behavioral: ELEVATE-S — ELEVATE-S uses implementation strategies to support clinicians (support clinicians by revising professional roles to enable point of care tobacco treatment with a team are approach and support clinicians by providing clinical decision support tools) and implementation strategies to support patients with chronic care model-informed self-management support (patient centered flexible goals and patient-generated health data).
  Arms: Electronic health record-enabled evidence-based tobacco treatment-Support (ELEVATE-S)

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of two different informatics-enabled implementation strategies on increasing tobacco treatment and improving smoking cessation rates for cancer control and prevention. This will be done via a two-arm pragmatic cluster randomized trial (CRT) to test the effectiveness of nudges to change (ELEVATE-S) vs. quit-focused usual care (ELEVATE) in increasing tobacco treatment (use of medication, brief advice, or referral to external counseling) and smoking cessation.

ELIGIBILITY:
Eligibility Criteria:

* Be receiving care at a participating clinic
* Report current tobacco use (assessed by the rooming staff during the index visit)
* Have a completed appointment with a participating clinic
* Be an adult (at least 18 years old).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient receipt of tobacco use treatment, i.e. Tobacco use treatment (TUT) Reach | Up to 6 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment (either medication or behavioral intervention (brief advice or referral to counseling)).

SECONDARY OUTCOMES:
Patient receipt of tobacco use treatment - behavioral intervention. | Up to 6 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment behavioral intervention (brief advice or referral to counseling).
Patient receipt of tobacco use treatment - medication. | Up to 6 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment medication.
Patient smoking abstinence | Up to 6 months post-enrollment
  This will be quantified by the proportion of patients who smoke with EHR-documented smoking abstinence

OTHER OUTCOMES:
Patient receipt of tobacco use treatment, i.e. Tobacco use treatment (TUT) Reach | Up to 12 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment (either medication or behavioral intervention (brief advice or referral to counseling).
Patient receipt of tobacco use treatment - behavioral intervention. | Up to 12 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment behavioral intervention (brief advice or referral to counseling).
Patient receipt of tobacco use treatment - medication. | Up to 12 months post-enrollment
  This will be quantified by the proportion of enrolled patients who receive tobacco use treatment medication.
Patient smoking abstinence | Up to 12 months post-enrollment
  This will be quantified by the proportion of patients who smoke with EHR-documented smoking abstinence
Patient bioverified smoking | Up to 12 months post-enrollment
  This will be quantified by the proportion of patients who smoke with bioverified point-prevalent abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiun Chen, M.D., MPH, ScD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu